CLINICAL TRIAL: NCT01715844
Title: L-Citrulline Supplementation Pilot Study for Overweight Late Onset Asthmatics
Acronym: SANDIA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Fernando Holguin, Assistant Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: L-citrulline Asthma
Record Dates: First submitted 2012-10-16; First posted 2012-10-29 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: L-citrulline; ADMA; Asthma; Obesity
MeSH Terms: conditions — Asthma; Obesity | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-citrulline (Active Comparator): 3-gr/day of L-citrulline effervescent powder mix
  Interventions: Dietary Supplement: L-citrulline
- Placebo (Placebo Comparator): 3 gr of Placebo/day matching L-citrulline effervescent powder
  Interventions: Dietary Supplement: L-citrulline

INTERVENTIONS:
Dietary Supplement: L-citrulline — Patients will take 3-gr of L-citrulline/day for 7 days
  Other Names: L-citrulline 3 gr efervescent powder

SUMMARY:
In people who develop asthma after the age of 12 and who are also overweigh, there can be an increased burden of asthma symptoms, more flare-ups, and poorly-controlled asthma when compared to normal weight asthmatics. Certain factors are more abundant in the blood of individuals who are obese. One such factor is derived from the metabolism of an amino acid found in your diet, which is known as L-arginine (Amino acids are most commonly known as the building blocks of proteins, the same as the proteins found in food). This factor is called asymmetric dimethylarginine or ADMA. The balance of L-arginine to ADMA may be important to the health of subjects with asthma. The balance between L-arginine and ADMA plays an important role in producing nitric oxide (NO) in the airways. NO is normally produced in the lung and plays a major role in maintaining airways open and functioning normally. Our research has shown that in subjects with asthma who are overweight and developed asthma later in life, the combination of low L-arginine and high ADMA, may lead to lower NO levels. We are asking participants in this study to take L-citrulline, which is converted to L-arginine by your body, as a supplement for a period of one week. We anticipate that L-citrulline will restore NO levels in the airways, by increasing the ratio of L-arginine to ADMA

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, 18-75 yrs old, from all racial/ethnic backgrounds
* Diagnosis of asthma for >1 yr
* BMI ≥ 30
* Baseline pre-bronchodilator FEV1 between 60 and 90% predicted with a 12% or greater bronchodilator response to 4 puffs of albuterol
* Smoking history <20 pack years and no smoking in the last year
* Able to identify age of asthma onset

Exclusion Criteria:

* Respiratory tract infection within the last 4 weeks;
* Oral CS burst within the last 4 weeks or regular systemic CS use
* Hospitalization within the last 3 months
* ER visit within the 4 weeks
* Significant or uncontrolled concomitant medical illness including (but not limited to) heart disease, cancer, diabetes
* Current smoking or within the previous 12 months
* Current use of statins for the past 30 days (Statins lower ADMA levels)
* Pregnancy
* Intolerance or allergy to L-arginine or L-citrulline
* Phosphodiesterase inhibitors
* Taking oral nitrates

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09-07 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Exhaled nitric oxide | 1 week
  Patients will be randomized to 1 week of 3 g of L-citrulline/day vs matching placebo, The outcome is the pre to post intervention change in exhaled NO

SECONDARY OUTCOMES:
Sputum and plasma L-arginine/ADMA levels | 1 week
  This outcome compares the pre to post L-citrulline supplementation changes in sputum and plasma L-arginine/ADMA

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Holguin, MD MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- Asthma Institute, University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Holguin F, Grasemann H, Sharma S, Winnica D, Wasil K, Smith V, Cruse MH, Perez N, Coleman E, Scialla TJ, Que LG. L-Citrulline increases nitric oxide and improves control in obese asthmatics. JCI Insight. 2019 Dec 19;4(24):e131733. doi: 10.1172/jci.insight.131733. PMID 31714895